CLINICAL TRIAL: NCT03199989
Title: Efficacy of Postoperative Adjuvant Chemotherapy for Stage II Colon Cancer With High Risk Factors(EPAC1)
Acronym: EPAC1
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Peking Union Medical College Hospital (Other); Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Aiwen Wu, M.D. PH.D. Chief, Unit III & Ostomy Service, Gastrointestinal Cancer Center, Peking University Cancer Hospital & Institute, Peking University Cancer Hospital & Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKUCH-C01
Record Dates: First submitted 2017-06-04; First posted 2017-06-27 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Adjuvant Chemotherapy
Keywords: colon cancer; adjuvant chemotherapy; high risk
MeSH Terms: conditions — Colonic Neoplasms | interventions — Observation

STUDY DESIGN:
Intervention Model Description: a prospertive randomized clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- adjuvant chemotherapy group (Active Comparator): patients enrolled int the adjuvant chemotherapy group will receive adjuvant chemotherapy[CapeOX（Capecitabine+Oxaliplatin）] by the current guidelines
  Interventions: Drug: CapeOX（Capecitabine+Oxaliplatin）
- observation group (Experimental): patients enrolled int the adjuvant chemotherapy group will not receive adjuvant chemotherapy just for observation
  Interventions: Other: Observation

INTERVENTIONS:
Drug: CapeOX（Capecitabine+Oxaliplatin） — Patients enrolled in the chemotherapy group would receive postoperative chemotherapy CapeOX（Capecitabine+Oxaliplatin）for 6 months
  Arms: adjuvant chemotherapy group
Other: Observation — Patients enrolled in the observation group would not receive any chemotherapy drugs just for observation
  Arms: observation group

SUMMARY:
The purpose of this study is to design a prospective randomized clinical trial to explore whether postoperative adjuvant chemotherapy may provide survival benefit for stage II colon cancer patients with high risk factors.Therefore the investigators can provide high level clinical evidence of indications for patients with colon cancer with stage II colon cancer.

DETAILED DESCRIPTION:
The most controversial of adjuvant chemotherapy for colon cancer is whether stage II colon cancer should receive adjuvant chemotherapy or not. Because of the absolute little benefit of adjuvant chemotherapy after curative resection of stage II colon cancer，NCCN and ESMO guidelines do not recommend routine adjuvant chemotherapy for patients with stage II colon cancer unless combined with high risk factors.

Currently，most studies about stage II colon cancer with high risk factors were retrospective. Some suggested that patients with stage II colon cancer can benefit from adjuvant chemotherapy, however, more got the negative conclusions.

The study was designed as a multicenter, prospective, randomized, controlled trial.Patients who agreed to participate in the study would be randomly assigned to a treatment group of adjuvant chemotherapy or observation with 50% chance by a central randomization system determined by the computer program.

After a follow up of at least 3 years, the disease free survival of the two groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 to 75 years;
2. pathologically confirmed adenocarcinoma of the colon
3. after curative resection pathological stage was T3-4N0M0;
4. with at least one of the following factors:

   1. T4 staging
   2. lymph nodes number less than 12
   3. poor differentiation (except MSI-H)
   4. LVI or PNI
   5. obstruction or perforation
   6. Elevated preoperative serum CEA
5. ECOG Performance status 0-1
6. no evidence of distant metastases
7. no preoperative chemotherapy or chemoradiation therapy
8. ANC > 1.5 cells/mm3, HGB > 10.0 g/dL, PLT > 100,000/mm3, total bilirubin ≤ 1.5 xULN, AST≤ 3 x ULN, ALT ≤ 3 x ULN.
9. Patients must read, agree to, and sign a statement of Informed Consent prior to participation in this study.

Exclusion Criteria:

1. combined with other cancer
2. Creatinine level greater than 1.5 times the upper limit of normal.
3. Patients who have received preoperative chemotherapy or chemoradiotherapy.
4. Patients with a history of a prior malignancy within the past 5 years.
5. Women who are pregnant or breast-feeding.
6. patients may not complete the whole schedule of chemotherapy
7. Patients with any other concurrent medical or psychiatric condition or disease which would make them inappropriate candidates for entry into this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1254 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival | At least 3 years after the last patient enrolled
  Disease free survival was defined as the duration after local recurrence or metastasis were found after surgery. Metastasis of any distant organs such as liver, lung, ovary，bone and peritoneum were defined by CT.

SECONDARY OUTCOMES:
3-year overall survival | At least 3 years after the last patient enrolled
  Overall survival was defined as the duration from randomization to death from any cause
Rate of metastasis | At least 3 years after the last patient enrolled
  Rate of metastasis in different groups
Relationship between high risk factors and survival | At least 3 years after the last patient enrolled
  All the high risk factors enrolled in this study will be analyzed one by one to investigate the relationship between high risk factors and survival.
Major adverse events | At least 1 years after the last patient enrolled
  Toxic reaction in the chemotherapy group.Adverse events will be graded using the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Aiwen Wu, M.D., Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing cancer hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No